CLINICAL TRIAL: NCT06970717
Title: Programmable Smart Watch for Remote Pre-habilitation/Rehabilitation Monitoring
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024/4048
Record Dates: First submitted 2025-03-03; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-02

CONDITIONS: Rehabilitation Exercise

STUDY DESIGN:
Intervention Model Description: 20 healthy volunteers will be recruited via hospital posters and email. Volunteers will receive a smartwatch and tablet for one week.
  After consent, they'll be shown 7 standard cancer prehabilitation exercises (Squat Chop, Ice-skater, Dig and Flex, Tap and Punch, March and Twist, Cross Punch, Sit-to-stand) demonstrated by a team member, and given exercise videos (via tablet/QR code).
  The 20-minute exercise session will be supervised, with posture correction and home exercise tips.
  Smartwatch data will be captured during the supervised session. Volunteers will then wear the watch and follow the videos for 5 days, exercising at their convenience, logging activity, and transmitting data to the tablet. No personal data will be entered.
  Finally, volunteers return the devices and complete a usability survey. Data will be compared against logs to assess accuracy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention arm (Experimental)
  Interventions: Device: M5Stick Programmable watch

INTERVENTIONS:
Device: M5Stick Programmable watch — This smart watch is fashioned using a M5StickC, an IOT platform which is programmable and allows us to measure specific exercises.

SUMMARY:
The purpose of this research study is to validate the M5Stick Programmable watch as a prototype to monitor specific prehabilitation exercises and to monitor the frequency of exercises and the number of repetitions the subject makes in a home setting.

DETAILED DESCRIPTION:
Background of study Locally, a digital platform, the Cancer prehabilitation exercise diary was developed by Singhealth Marcom with Changi General Hospital (CGH) to support a home-based cancer prehabilitation program complete with exercise videos and reminders. The disadvantage of home-based or remote rehabilitation and prehabilitation compared to a centre-based treatment is that of a lack of monitoring and reduced compliance. In the CGH home-based model of cancer prehabilitation, compliance is monitored by verbal confirmation over a telephone call made by the cancer prehabilitation coordinator at mid-point of the course, and then with verbal checking with the patient at the end of the prehabilitation program, at the pre-op visit.

With the direction of increased digitalization for healthcare of the future, there is a desire to develop a smart watch that allows for the monitoring of the frequency and accuracy of the exercises prescribed asynchronously. A summary of the patient's exercise frequency/intensity and accuracy can be gathered from the app on the accompanying tablet.

This prototype will be developed through collaboration with the Eastern General Hospital {EGH) Engineering department. There is currently no product on the market that will be customizable for the specific calisthenic and plyometric exercises that are part of the cancer prehabilitation exercise videos.

Specific aims of this study This study aims to validate the MSStick Programmable watch as a prototype to monitor specific prehabilitation exercises and to monitor the frequency of exercises and the number of repetitions the subject makes in a home setting.

Hypothesis of this study The hypothesis is that the MSStick Programmable watch is able to monitor the specific prehabilitation exercises performed in a home-setting by healthy volunteers, and is able to distinguish its frequency and number of repetitions

Importance of this study This project aims to develop a programmable smartwatch for remote prehabilitation/rehabilitation monitoring. We address the limitations of current home-based programs by enabling asynchronous monitoring of exercise frequency, accuracy, and intensity. The smartwatch utilizes a 6-axis Inertial Measurement Unit (IMU) to differentiate specific exercises and measure workout intensity.

Prototype validation will involve 20 healthy volunteers performing 7 pre-defined exercises. The smartwatch will capture data and compare it with volunteer logs to assess Its ability to capture specific and accurate data.

Based on the findings, further refinement of the programming, prototype, and work processes may be necessary. Future steps include cloud-based data transmission, commercialization, and validation with specific patient populations. This smartwatch has the potential to be an important tool for scaling up telerehabilitation and teleprehabilitation programs.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-60
2. Not on follow up for chronic diseases
3. Willing to perform exercises daily x 5 days
4. Able to handle simple technology eg. smart phone

Exclusion Criteria:

1. Pregnant women
2. Active joint pains and any other musculoskeletal issues
3. Heart conditions or balance issues

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Exercise Compliance | Over 1 week
  Measure if the exercises were performed as prescribed, based on the number of repetitions, the number of sets of exercises and the frequency of exercise

SECONDARY OUTCOMES:
Usability | over 1 week
  A survey using the mhealth usability questionaire, with 18 questions, each question with scores of 1 to 7, 7 being fully agree and 1 fully disagree.

OTHER OUTCOMES:
Technical reliability | over 1 week
  To measure if the device was able to synchronise with the app

CONTACTS AND LOCATIONS:
Locations (1):
- Changi General Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Data is protected under the SingHealth Data Protection Policy which is compliant to the Singapore Personal Data Protection Act 2012